CLINICAL TRIAL: NCT05421273
Title: Effects of Active Versus Passive Recharge Burst Spinal Cord Stimulation on Pain Experience in Persistent Spinal Pain Syndrome Type 2: a Multicenter Randomized Trial (BURST-RAP Study)
Acronym: BURST-RAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL75451.091.020
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Persistent Spinal Pain Syndrome Type 2; Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active recharge burst stimulation (Experimental)
  Interventions: Device: Spinal cord stimulation using active recharge burst stimulation
- Passive recharge burst stimulation (Experimental)
  Interventions: Device: Spinal cord stimulation using passive recharge burst stimulation

INTERVENTIONS:
Device: Spinal cord stimulation using passive recharge burst stimulation — Passive recharge burst is marked by a recharge pattern that passively compensates for charge differences.
  Arms: Passive recharge burst stimulation
Device: Spinal cord stimulation using active recharge burst stimulation — Active recharge burst is characterized by negative pulses that directly compensate for charge differences.
  Arms: Active recharge burst stimulation

SUMMARY:
Spinal cord stimulation (SCS) has shown to be an effective treatment for patients with persistent spinal pain syndrome Type 2 (PSPS Type 2). The method used to deliver electrical charge in SCS is important. One such method is burst stimulation. Two variations of burst waveforms are currently in use: one that employs active recharge and one that uses passive recharge. It is still unknown if there are clinical differences between active recharge and passive recharge burst SCS. To date, no clinical studies have been performed that directly compared these two burst stimulation waveforms. The objective of this Randomized Clinical Trial (RCT) is to assess and compare effect of passive recharge burst SCS with active recharge burst SCS on pain relief and motivational-emotional facets of pain

DETAILED DESCRIPTION:
This multicenter randomized clinical trial will take place in 6 Dutch hospitals: the Rijnstate Hospital (Arnhem), Bravis Hospital (Roosendaal), Elizabeth TweeSteden Hospital (Tilburg), Diakonessen Hospital (Utrecht), Alrijne Hospital (Leiden) and the Amsterdam University Medical Hospitals A-UMC). PSPS Type II2 patients (n=96) will be randomized into a group receiving either active or passive recharge burst. Following a successful trial period, patients are permanently implanted. Patients complete the pain catastrophizing score (PCS) (primary outcome at 6 months), numeric pain rating scale (NRS), patient vigilance and awareness questionnaire (PVAQ), hospital anxiety and depression scale (HADS), quality of life (EQ-5D), Oswestery disability index (ODI), patient global impression of change (PGIC) and painDETECT questionnaires (secondary outcomes) at baseline, after trial, 1, 3, 6 and 12 months following implantation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 70 years of age
* At least moderate level of catastrophizing as measured with the Pain catastrophizing scale (PCS) of at least 20 at first visit of the pain clinic.
* Chronic pain diagnoses as PSPS Type 2 of at least 6 months
* Neurologic exam without marked motor deficit.
* LBP and/or leg pain intensity should be 5 or higher measured with the 11-box NRS 0-10
* Meets all the inclusion criteria for the implantation of a neurostimulation system as typically utilized in the study center. PM: depression is not an exclusion criteria
* Subject has been screened by a multi-disciplinary panel including a psychologist and deemed suitable for implantation
* Subject is able and willing to comply with the follow-up schedule and protocol
* Subject is able to provide written informed consent

Exclusion Criteria:

* Female subject of childbearing potential is pregnant/nursing or plans to become pregnant during the course of the study
* Escalating or changing pain condition within the past month as evidenced by investigator examination
* BMI ≥35
* "Subject has had injection therapy or radiofrequency treatment for their low back pain (LBP) or leg pain within the past 3 months"
* Subject currently has an active implantable device including ICD, pacemaker, spinal cord stimulator or intrathecal drug pump
* Subject is unable to operate the device
* Severe spinal column degeneration likely to cause technical problems with neuromodulation, to be assessed by the treating physician
* Previous Neurostimulation therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain catastrophizing score | 6 months

SECONDARY OUTCOMES:
Numeric pain rating scale | 3, 6, 12 months
Patient vigilance and awareness questionnaire | 3, 6, 12 months
Hospital anxiety and depression scale | 3, 6, 12 months
EQ-5D questionnaire | 3, 6, 12 months
  Quality of life questionnaire
Oswestery disability index | 3, 6, 12 months
Patient global impression of change | 3, 6, 12 months
PainDETECT questionnaire | 3, 6, 12 months
  Characterisation of neuropathic pain components
Mean charge per second used | 3, 6, 12 months
  Measures the amount of electrical charge used
Mean charge per hour used | 3, 6, 12 months
  Measures the amount of electrical charge used

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Bravis Hospital, Roosendaal, North Brabant
  - Elizabeth TweeSteden Hospital, Tilburg, North Brabant
  - Amsterdam University Medical Hospitals A-UMC, Amsterdam, North Holland
  - Alrijne Hospital, Leiderdorp, South Holland
  - Diakonessen Hospital, Zeist, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mons MR, Edelbroek C, Zuidema X, Burger K, Elzinga L, de Vries J, van Kuijk S, Joosten EA, Kallewaard JW. Study protocol: Effects of active versus passive recharge burst spinal cord stimulation on pain experience in persistent spinal pain syndrome type 2: a multicentre randomized trial (BURST-RAP study). Trials. 2022 Sep 5;23(1):749. doi: 10.1186/s13063-022-06637-7. PMID 36064598